CLINICAL TRIAL: NCT04833101
Title: Safety and Immunogenicity of a Heterologous Immunization of Recombinant COVID-19 Vaccine (Ad5 Vector) and RBD-based Protein Subunit Vaccine Against COVID-19 in Chinese Healthy Population
Brief Title: Study on Heterologous Prime-boost of Recombinant COVID-19 Vaccine (Ad5 Vector) and RBD-based Protein Subunit Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT115
Record Dates: First submitted 2021-04-03; First posted 2021-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2 Vaccine; Recombinant Ad5 Vector; Subunit Vaccine; Safety; Immunogenicity
MeSH Terms: conditions — COVID-19 | interventions — Ad5-nCoV vaccine; ZF2001 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- "0-28 days" vaccine group (Experimental): One dose of recombinant Ad5 vectored COVID-19 vaccine on day 0, the second dose of subunit vaccine (ZF2001) against COVID-19 on day 28, and a third of subunit vaccine (ZF2001) against COVID-19 on month 4.
  Interventions: Biological: recombinant Ad5 vectored COVID-19 vaccine; Biological: RBD-based protein subunit vaccine (ZF2001) against COVID-19
- "0-28 days" placebo group (Placebo Comparator): One dose of recombinant Ad5 vectored COVID-19 vaccine on day 0, the second dose of a commercial influenza vaccine on day 28, a third of subunit vaccine (ZF2001) against COVID-19 on month 4.
  Interventions: Biological: recombinant Ad5 vectored COVID-19 vaccine; Biological: RBD-based protein subunit vaccine (ZF2001) against COVID-19; Biological: trivalent split influenza vaccine
- "0-56 days" vaccine group (Experimental): One dose of recombinant Ad5 vectored COVID-19 vaccine on day 0, the second dose of subunit vaccine (ZF2001) against COVID-19 on day 56, a third of subunit vaccine (ZF2001) against COVID-19 on month 4.
  Interventions: Biological: recombinant Ad5 vectored COVID-19 vaccine; Biological: RBD-based protein subunit vaccine (ZF2001) against COVID-19
- "0-56 days" placebo group (Placebo Comparator): One dose of recombinant Ad5 vectored COVID-19 vaccine on day 0, the second dose of a commercial influenza vaccine on day 56, a third of subunit vaccine (ZF2001) against COVID-19 on month 4.
  Interventions: Biological: recombinant Ad5 vectored COVID-19 vaccine; Biological: RBD-based protein subunit vaccine (ZF2001) against COVID-19; Biological: trivalent split influenza vaccine

INTERVENTIONS:
Biological: recombinant Ad5 vectored COVID-19 vaccine — This vaccine contains 5×10^10 virus particles of recombinant replication defective human type-5 adenovirus expressing SARS-CoV-2 S protein, which is produced by CanSino Biologics Inc. It is a liquid dosage form, 0.5 ml / bottle.
  Other Names: Ad5-nCoV
Biological: RBD-based protein subunit vaccine (ZF2001) against COVID-19 — This is a recombinant tandem-repeat dimeric RBD-based protein subunit vaccine (ZF2001) against COVID-19, made by using CHO cell, 25μg/dose, produced by Anhui Zhifei Longcom Biopharmaceutical Co.,Ltd.
  Other Names: ZF2001 vaccine
Biological: trivalent split influenza vaccine — This vaccine contains 15 μ g H1NI, 15 μ g H3N2 and 15 μ g B-series hemagglutinin, produced by Dalian Aleph Biomedical Co., Ltd.It is a liquid dosage form, 0.5 ml / bottle.
  Arms: "0-28 days" placebo group; "0-56 days" placebo group

SUMMARY:
This is a randomized, observer-blind, placebo-controlled study, for evaluation of safety and immunogenicity of heterologous prime-boost immunization of recombinant COVID-19 vaccine (adenovirus type-5 vector) and RBD-based protein subunit vaccine (ZF2001) against COVID-19 in Chinese healthy population. 120 healthy subjects aged over 18 years of age who have been vaccinated with recombinant adenovirus type-5 vectored vaccine will be recruited in this study. Of them, 60 subjects will be enrolled in the "0-28 days" regimen and other 60 will be enrolled in "0-56 days" regimen. Subjects, 30 of them are 18-59 years old and 30 are 60 years old and above in each regimen will be randomly vaccinated with the second dose of subunit vaccine(ZF2001) against COVID-19 or a commercial influenza vaccine in a ratio of 2:1. They will then be vaccinated with the third dose of ZF2001 on month 4 after the second dose. The occurrence of adverse events within 28 days and serious adverse events within 6 months after the last vaccination will be observed. In addition, blood samples will be collected on day 0 before the second vaccination, day 14, 28 after the second vaccination and day 14, month 6 after third vaccination to test serum antibody levels and to profile the immune cells' subgroups and germlines. Each subject will remain in this study for approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* The subjects ≥ 18 years old who has completed one dose of recombinant Ad5 vectored COVID-19 vaccine.
* The subjects can provide with informed consent and sign informed consent form (ICF).
* The subjects are able to and willing to comply with the requirements of the clinical trial program and can complete the 6-month follow-up of the study.
* Axillary temperature ≤ 37.0 ℃
* Individuals who are in good health condition at the time of entry into the trial as determined by medical history, physical examination and clinical judgment of the investigator and meet the requirements of these products immunization.

Exclusion Criteria:

* have a medical history or family history of convulsion, epilepsy, encephalopathy and psychosis.
* be allergic to any component of the research vaccines, or used to have a history of hypersensitivity or serious reactions to vaccination.
* Women with positive urine pregnancy test, pregnant or breast-feeding, or have a pregnancy plan within six months.
* have acute febrile diseases and infectious diseases.
* have severe chronic diseases or condition in progress cannot be smoothly controlled, such as asthma, diabetes, thyroid disease
* Congenital or acquired angioedema / neuroedema.
* have the history of urticaria 1 year before receiving the trial vaccine.
* have asplenia or functional asplenia.
* have thrombocytopenia or other coagulation disorders (which may cause contraindications for intramuscular injection).
* have the history of immunosuppressive therapy, anti allergy therapy, cytotoxic therapy or inhaled corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis, and acute corticosteroid therapy without dermatitis) over the past 6 months.
* have received blood products within 4 months before injection of trial vaccines.
* have received another investigational product within one month before injection of trial vaccine.
* have received attenuated vaccine within 1 month before injection of trial vaccine except the recombinant Ad5 vectored COVID-19 vaccine.
* have received subunit or inactivated vaccine within 14 days before the vaccination with trial vaccine.
* under anti tuberculosis treatment.
* not be able to follow the protocol, or not be able to understand the informed consent according to the researcher's judgment, due to various medical, psychological, social or other conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited adverse events within 7 days after vaccination. | Within 7 days after vaccination
  Incidence of solicited adverse events within 7 days after vaccination.
GMT of neutralizing antibodies against live SARS-CoV-2 virus at Day 14 after the booster vaccination. | At Day 14 after the booster vaccination
  GMT of neutralizing antibodies against live SARS-CoV-2 virus at Day 14 after the booster vaccination.

SECONDARY OUTCOMES:
Incidence of adverse reactions within 28 days after vaccination. | Within 28 days after vaccination
  Incidence of adverse reactions within 28 days after vaccination.
Incidence of adverse events within 28 days after vaccination. | Within 28 days after vaccination.
  Incidence of adverse events within 28 days after vaccination.
Incidence of unsolicited AE within 28 days after vaccination. | Within 28 days after vaccination.
  Incidence of unsolicited adverse events within 28 days after vaccination.
Incidence of serious adverse events(SAE) from the first dose to the 6 months after completing the last dose of vaccination. | From the first dose to the 6 months after completing the last dose of vaccination.
  Incidence of serious adverse events(SAE) from the first dose to the 6 months after completing the last dose of vaccination.
GMT of binding antibodies against SARS-CoV-2 S and RBD protein measured by ELISA at day 14, day 28 after the second vaccination, and day 14, month 6 after the third vaccination. | at day 14, day 28 after the second vaccination, and day 14, month 6 after the third vaccination.
  GMT of binding antibodies against SARS-CoV-2 S and RBD protein measured by ELISA at day 14, day 28 after the second vaccination, and day 14, month 6 after the third vaccination.
Proportion of the participants with at least a four-fold increase of the binding antibodies against SARS-CoV-2 S and RBD protein at day 14, day 28 after the second vaccination, and day 14, month 6 after the third vaccination. | at day 14, day 28 after the second vaccination, and day 14, month 6 after the third vaccination.
  Proportion of the participants with at least a four-fold increase of the binding antibodies against SARS-CoV-2 S and RBD protein at day 14, day 28 after the second vaccination, and day 14, month 6 after the third vaccination.
Fold increase of binding antibodies against SARS-CoV-2 S and RBD protein at day 14, day 28 after the second vaccination, and day 14, month 6 after the third vaccination. | at day 14, day 28 after the second vaccination, and day 14, month 6 after the third vaccination.
  Fold increase of binding antibodies against SARS-CoV-2 S and RBD protein measured by ELISA, as compared to baseline, at day 14, day 28 after the second vaccination, and day 14, month 6 after the third vaccination.
GMT of neutralizing antibodies against live SARS-CoV-2 virus at day 28 after the second vaccination, and day 14, month 6 after the third vaccination | at day 28 after the second vaccination, and day 14, month 6 after the third vaccination
  GMT of neutralizing antibodies against live SARS-CoV-2 virus at day 28 after the second vaccination, and day 14, month 6 after the third vaccination
Proportion of the participants with at least a four-fold increase of neutralizing antibodies against live SARS-CoV-2 virus at day 14, day 28 after the second vaccination, and day 14, month 6 after the third vaccination. | at day 14, day 28 after the second vaccination, and day 14, month 6 after the third vaccination.
  Proportion of the participants with at least a four-fold increase of neutralizing antibodies against live SARS-CoV-2 virus, as compared to baseline, at day 28 after the second vaccination, and day 14, month 6 after the third vaccination.
Fold increase of neutralizing antibodies against live SARS-CoV-2 virus at day 14, day 28 after the second vaccination and day 14, month 6 after the third vaccination. | at day 14, day 28 after the second vaccination and day 14, month 6 after the third vaccination.
  Fold increase of neutralizing antibodies against live SARS-CoV-2 virus, as compared to baseline, at day 14, day 28 after the second vaccination and day 14, month 6 after the third vaccination.

OTHER OUTCOMES:
Types of binding antibodies IgG against SARS-CoV-2 S protein at day 14, day 28 after the second vaccination and day 14, month 6 after the third vaccination. | at day 14, day 28 after the second vaccination and day 14, month 6 after the third vaccination.
  Types of binding antibodies IgG against SARS-CoV-2 S protein at day 14, day 28 after the second vaccination and day 14, month 6 after the third vaccination.
Cross neutralizing of the antibodies to variants of SARS-CoV-2 measured by pseudovirus neutralization test at Day 28 after the booster vaccination. | At Day 28 after the booster vaccination.
  Cross neutralizing of the antibodies to variants of SARS-CoV-2 measured by pseudovirus neutralization test at Day 28 after the booster vaccination.
The immune cells' subgroups and germlines at Day 28 after vaccination. | At Day 28 after vaccination.
  The immune cells', such as B cells and T cells, subgroups and germlines at Day 28 after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Xin Li, PhD, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be available for request 1 month after the completion of the study
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 1 month to 1 year after the completion of the study
Access Criteria: Researchers who provide a scientifically sound proposal will be allowed access to the individual participant data.These proposals will be reviewed and approved by the sponsor, investigator, and collaborators on the basis of scientific merit. To gain access, data requesters will need to sign a data access agreement.

REFERENCES:
- [Derived] Jin P, Guo X, Chen W, Ma S, Pan H, Dai L, Du P, Wang L, Jin L, Chen Y, Shi F, Liu J, Xu X, Zhang Y, Gao GF, Chen C, Feng J, Li J, Zhu F. Safety and immunogenicity of heterologous boost immunization with an adenovirus type-5-vectored and protein-subunit-based COVID-19 vaccine (Convidecia/ZF2001): A randomized, observer-blinded, placebo-controlled trial. PLoS Med. 2022 May 26;19(5):e1003953. doi: 10.1371/journal.pmed.1003953. eCollection 2022 May. PMID 35617368